CLINICAL TRIAL: NCT03144440
Title: Real World Experience of Chronic Hepatitis C Treatment in Israeli Patients With Advanced Liver Fibrosis With Fixed Dose Combination (FDC) Grazoprevir (100 mg)/Elbasvir (50mg) (Zepatier) ± Ribavirin: A Retrospective Multicenter Cohort Study
Brief Title: Real World Experience of Chronic Hepatitis C (CHC) Treatment in Israel
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eli Zuckerman, Prof. Eli Zuckerman, Carmel Medical Center
Other Study IDs: CMC-16-0096-CTIL
Record Dates: First submitted 2017-03-14; First posted 2017-05-08 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis C
Keywords: ZEPATIER
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective:

1. To estimate the effectiveness of treatment with FDC of Zepatier with or without ribavirin in Israeli patients with CHC and advanced fibrosis in real life setting.

Secondary objective:

1. To estimate the safety and tolerability of treatment with FDC of Zepatier with or without ribavirin in real life setting in Israeli patients with CHC and advanced disease.

Hypotheses:

Effectiveness and tolerability of treatment with FDC of Zepatier with or without ribavirin in Israeli patients with CHC and advanced fibrosis will be similar to that demonstrated in phase 3 clinical trials.

DETAILED DESCRIPTION:
The following data will be collected:

Demographics information: age, gender, race, country of birth (COB). Data on liver and virological characteristics: Hepatitis C virus(HCV) genotype, fibrosis stage (F0-4), technology of fibrosis assessment (fibroscan, fibrotest, elastography, biopsy), , cirrhosis (y/n), presence of portal hypertension: esophageal varices, ascites, hepatic encephalopathy, history of decompensation, liver transplantation (y/n).

Previous anti-viral treatment: PR- Peg-Riba (relapse, partial/null responder, unknown response), direct anti-viral agents (DDAs): Protease Inhibitors (PI) (Bocepravir,Telepravir, Simepravir), Sofosbuvir (SOF), NS5A (Ledipasvir, Daclatasvir), NS5B.

Co-morbidities: BMI, Diabetes Mellitus, HIV-co infection, HBV-co infection, alcohol abuse, CKD (Chronic kidney disease)/renal failure, cardiovascular disease, inherited blood disorders, pre/post-transplant (liver/kidney) Concomitant medication (drug-drug interactions): antiacids (Proton pump inhibitors,H2-blockers), statins,beta-blockers, oral contraceptives, anti hypertensive, Anti retrovirals for HIV, etc.

Base line and end-of treatment parameters: White blood cells(WBC), Hemoglobin (HB), Platelates (PLT), Alanine transferase (ALT), Aspartate transaminase (AST), Alpha phetoprotein (ALP), Gamma glutamyl transferase (GGT), albumin, bilirubin, Protrombin time (PT)/INR, LDL-C, IL28 (if available), Model for end stage liver disease (MELD) score, Child pugh (CPT) score/class, viral load and virological response: HCV ribonucleic acid (RNA) at week 4 and 8 (if available), and sustained virological response (SVR) 12 and SVR24.

Data on virological breakthrough and relapse will be also collected and if possible to check resistance associated variants (RAVs).

Data on treatment safety: any adverse event (AE), serious adverse event (SAE), AE which led to early discontinuation of treatment; decompensation event (ascites, hepatic encephalopathy, bleeding esophageal varices,) liver failure, liver transplantation and death.

Primary variable The proportion of patients achieving SVR12 (HCV RNA <15 IU/mL at follow-up week 12; 12 weeks after the last actual dose of the Zepatier).

The Full Analysis Set will include all patients who received ≥1 dose of Zepatier.

Secondary variables

* Cirrhosis/Fibrosis stage (F3, F4). Cirrhosis defined by liver biopsy (Metavir F4); transient elastography by Fibroscan tomography (TM) (>12.5 kPa); or FibroTest® or FibroSure® (>0.75 with APRI >2).
* Previous HCV anti-viral treatment
* Co-morbidities and concomitant medication
* Laboratory abnormalities; baseline and end of treatment (EoT) parameters
* Serious and non-serious adverse events occurring at any time during the treatment period, and other adverse events up until 14 days after cessation of treatment, will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients that treated with Zepatier after SVR results

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data collection from electronic patients' files from the different medical centers participating in the study will be performed after completion of treatment and follow-up period of up to 24 weeks post treatment (SVR).
  Data will be collected every 4 months (3 times a year) and analyzed in one center (Carmel Medical Center, Haifa, Israel).
  Study interim report will be provided twice per year (middle and end of each year)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with sustained virological response at week 12 (SVR12) [ Time Frame (for each patient): 12 weeks after the last dose of treatment ] | 12 weeks after the last dose of treatment
  SVR12 is defined as hepatitis c virus ribonucleic acid (HCV RNA) levels less than the lower limit of quantification 12 weeks after the last dose of treatment

SECONDARY OUTCOMES:
Safety of Elbasvir/Grazoprevir treatment against HCV infection in real-life conditions is reflected as the number of patients with clinical and biological adverse events occurring during the treatment . | 24 weeks
  Adverse event from the time when the decision is made to initiate treatment with Elbasvir/Grazoprevir until after the last dose

IPD SHARING:
Plan to Share IPD: No